CLINICAL TRIAL: NCT02245919
Title: A Primary Care Biopsychosocial Intervention (Back on Track) for Patients With Chronic Low Back Pain in Which Psychosocial Factors Moderately Influence Daily Life Functioning: a Pilot Study
Brief Title: Chronic Low Back Pain Rehabilitation in Primary Care: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Adelante, Centre of Expertise in Rehabilitation and Audiology (Other); The Province of Limburg (Unknown); CZ Fonds (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-3-024
Record Dates: First submitted 2014-09-16; First posted 2014-09-22 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2017-11

CONDITIONS: Chronic Low Back Pain
Keywords: Low Back Pain; Chronic Pain; Cognitive Behavioral Therapy; Primary Health Care; Physical Therapy
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Back on Track intervention (Experimental): A biopsychosocial primary care intervention based on multidisciplinary pain rehabilitation programs. The Back on Track intervention comprises 4 individual sessions and 8 group sessions.
  Interventions: Other: Back on Track intervention

INTERVENTIONS:
Other: Back on Track intervention — A biopsychosocial primary care intervention based on multidisciplinary pain rehabilitation programs. The Back on Track intervention comprises 4 individual sessions and 8 group sessions.

SUMMARY:
Up to now, only little research has been performed in tailoring treatment of patients with chronic low back pain (CLBP). It would be interesting to evaluate a biopsychosocial intervention in patients with a moderate to high level of disability and in whom the contributing role of psychosocial factors to this disability is mild to moderate (WPN3-). Nowadays, these patients receive cognitive behavioral-based treatments in multidisciplinary rehabilitation settings but might also benefit from treatments based on these multidisciplinary rehabilitation treatment principles when provided by specifically trained primary care physical therapists. Therefore, the aims of this pilot-study are to evaluate the feasibility of a specifically for primary care physiotherapist developed biopsychosocial intervention ("Back on Track" intervention) in WPN3- classified patients, and to evaluate whether this "Back on Track" intervention results in a significant improvement in functional disability in this subgroup of patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain; defined as pain between scapulae and gluteal region, whether or not with radiation towards one or both legs, present for at least three months.
* Presence of contributing social and psychological factors, however not complex (WPN3-classification).
* Age between 18 and 65 year
* Sufficient knowledge of the Dutch language
* Acceptance towards the biopsychosocial approach instead of biomedical approach

Exclusion Criteria:

* Chronic low back pain attributable to e.g. infection, tumour, osteoporosis, fracture, structural deformation, inflammatory process, radicular syndrome or cauda equina syndrome
* Pregnancy
* Any suspicion of an (underlying) psychiatric disease, for which psychiatric treatment is better suited, according to the expert opinion of the consultant in rehabilitation medicine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Quebec Back Pain Disability Scale (QBPDS) | Change in functional disability between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
  The QBPDS is a 20-itemed questionnaire designed to determine the individuals' functional disability level (ranging from 0-100). A higher score reflects higher disability.

SECONDARY OUTCOMES:
Credibility and Expectancy Questionnaire (CEQ) | Directly after the first treatment (in the first week of the intervention)
EuroQol-5D (EQ-5D) | Change in quality of life between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Hospital Anxiety and Depression Scale (HADS) | Change in anxiety and depression between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Pain Catastrophizing Scale (PCS) | Change in catastrophizing between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Numeric Rating Scale (NRS) | Change in catastrophizing between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Tampa Scale of Kinesiophobia (TSK) | Change in kinesiophobia between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Global Perceived Effect (GPE) | Global perceived effect at post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Trimbos and iMTA questionnaire on Costs associated with Psychiatric illness (TiC-P) | Medical consumption at pre-treatment (baseline), post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Social demographic questionnaire | pre-treatment (baseline)
Treatment satisfaction questionnaire | post-treatment (with an expected average of 8 weeks)
  This questionnaire will include questions about the patient's opinion regarding the intervention, the workbook, the consultant in rehabilitation medicine, the therapist(s), and the patient's perceived knowledge
Pain Self-Efficacy Questionnaire (PSEQ) | Change in self-efficacy between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Protocol adherence | All therapy sessions of the Back on Track intervention will be audio recorded (the intervention period of the trial will last approximately one year and 3 months)
  Physiotherapists will audio record all therapy sessions. A random sample will be assessed for protocol adherence using a modified version of the protocol used by Leeuw et al (2009). This protocol includes essential treatment elements and raters will judge whether these essential treatments elements are provided during the therapy or not. Adherence will be regarded sufficient in case a percentage of 70% of the required treatment elements are provided during the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan PJ Huijnen, Dr., Principal Investigator — Maastricht University Medical Center
Locations (4):
- Netherlands (4):
  - Fysiotherapie Abbink, Bunde, Limburg
  - Fysiohof, Maastricht, Limburg
  - ICM Fysio, Maastricht, Limburg
  - Fysiotherapie Breuers, Margraten, Limburg

REFERENCES:
- [Background] Vlaeyen JWS, Linton SJ. Fear-avoidance and its consequences in chronic musculoskeletal pain: a state of the art. Pain. 2000 Apr;85(3):317-332. doi: 10.1016/S0304-3959(99)00242-0. PMID 10781906
- [Background] Lindstrom I, Ohlund C, Eek C, Wallin L, Peterson LE, Fordyce WE, Nachemson AL. The effect of graded activity on patients with subacute low back pain: a randomized prospective clinical study with an operant-conditioning behavioral approach. Phys Ther. 1992 Apr;72(4):279-90; discussion 291-3. doi: 10.1093/ptj/72.4.279. PMID 1533941
- [Background] Leeuw M, Goossens MEJB, van Breukelen GJP, de Jong JR, Heuts PHTG, Smeets RJEM, Koke AJA, Vlaeyen JWS. Exposure in vivo versus operant graded activity in chronic low back pain patients: results of a randomized controlled trial. Pain. 2008 Aug 15;138(1):192-207. doi: 10.1016/j.pain.2007.12.009. Epub 2008 Feb 1. PMID 18242858
- [Background] Lamb SE, Hansen Z, Lall R, Castelnuovo E, Withers EJ, Nichols V, Potter R, Underwood MR; Back Skills Training Trial investigators. Group cognitive behavioural treatment for low-back pain in primary care: a randomised controlled trial and cost-effectiveness analysis. Lancet. 2010 Mar 13;375(9718):916-23. doi: 10.1016/S0140-6736(09)62164-4. Epub 2010 Feb 25. PMID 20189241
- [Background] Macedo LG, Smeets RJ, Maher CG, Latimer J, McAuley JH. Graded activity and graded exposure for persistent nonspecific low back pain: a systematic review. Phys Ther. 2010 Jun;90(6):860-79. doi: 10.2522/ptj.20090303. Epub 2010 Apr 15. PMID 20395306
- [Background] Brunner E, De Herdt A, Minguet P, Baldew SS, Probst M. Can cognitive behavioural therapy based strategies be integrated into physiotherapy for the prevention of chronic low back pain? A systematic review. Disabil Rehabil. 2013 Jan;35(1):1-10. doi: 10.3109/09638288.2012.683848. Epub 2012 May 21. PMID 22607157